CLINICAL TRIAL: NCT05130658
Title: Pilot Study to Improve Ambulation in Individuals With Traumatic Brain Injury (TBI) Using Virtual Reality -Based Treadmill Training
Brief Title: Study to Improve Ambulation in Individuals With TBI Using Virtual Reality -Based Treadmill Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-1125-20
Record Dates: First submitted 2021-09-16; First posted 2021-11-23 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- C-MILL training group (Experimental): The participants will be screened for the inclusion/exclusion criteria and consented during the first session. They will participate in two data collection sessions, one before the training and one after the training. The participants will undergo 10 training sessions. Individuals in the CTG will receive gait and balance training sessions with the virtual reality and auditory cues using C-MILL (such as walking on a pathway, obstacle avoidance, lateral balance etc.) to provide task specific training. C-Mill (Motekforce Link, Amsterdam, The Netherlands) is an instrumented treadmill that uses visual (on the screen as well on the treadmill) and acoustic cues for gait and balance training. The C-Mill allows for gait and balance adaptability strategy as it can provide obstacle avoidance environments, change in speed and various walking pathways in a safe and controlled environment.
  Interventions: Device: Virtual reality treadmill training
- Treadmill training group (TTG) (Active Comparator): The participants will be screened for the inclusion/exclusion criteria and consented during the first session. They will participate in two data collection sessions, one before the training and one after the training. The participants will undergo 10 training sessions. Individuals in TTG group will walk on the treadmill (C-MILL) or stand on the treadmill (C-MILL) with no visual or auditory cues.
  Interventions: Other: Treadmill Training
- Healthy Control (No Intervention): HCG will participate in up to four sessions. The participants will be screened for the inclusion/exclusion criteria and consented during the first session. They will participate in two data collection sessions and one C-MILL session.

INTERVENTIONS:
Device: Virtual reality treadmill training — C-Mill (Motekforce Link, Amsterdam, The Netherlands) is an instrumented treadmill that uses visual (on the screen as well on the treadmill) and acoustic cues for gait and balance training. The C-Mill allows for gait and balance adaptability strategy as it can provide obstacle avoidance environments, change in speed and various walking pathways in a safe and controlled environment.
  Other Names: C-MILL training, C-Mill (Motek, the Netherlands)
  Arms: C-MILL training group
Other: Treadmill Training — Conventional gait and balance training using treadmill.
  Arms: Treadmill training group (TTG)

SUMMARY:
The purpose of this research study is to test the effectiveness of virtual reality (VR) based treadmill training on walking ability. The study will also help to understand the changes in cognitive ability and brain activity as a result of VR-based treadmill training after a brain injury.

The study will include 3 groups: C-MILL training group (CTG), Treadmill training group (TTG), and healthy control group (HCG).

Individuals with brain injury will be randomly assigned to C-MILL training group, or Treadmill training group.

The CTG and TTG will participate in up to 13 sessions. The participants will be screened for the inclusion/exclusion criteria and consented during the first session. They will participate in two data collection sessions, one before the training and one after the training. The participants will undergo 10 training sessions. Individuals in the CTG will receive gait and balance training sessions with the virtual reality and auditory cues using C-MILL (such as walking on a pathway, obstacle avoidance, lateral balance etc.) to provide task specific training. C-Mill (Motekforce Link, Amsterdam, The Netherlands) is an instrumented treadmill that uses visual (on the screen as well on the treadmill) and acoustic cues for gait and balance training. The C-Mill allows for gait and balance adaptability strategy as it can provide obstacle avoidance environments, change in speed and various walking pathways in a safe and controlled environment.

Individuals in TTG group will walk on the treadmill (C-MILL) or stand on the treadmill (C-MILL) with no visual or auditory cues.

HCG will participate in up to four sessions. The participants will be screened for the inclusion/exclusion criteria and consented during the first session. They will participate in two data collection sessions and one C-MILLsession.

Each training session will last for 45 minutes. During the 45 minutes, the participants will perform the task for approximately 1 minute. Participants will be allowed as much rest as needed by them.

During the training all participants will wear the safety harness to protect from falling. In addition spotter will be present with the participants to prevent falls.

Data Collection:

Each participant's baseline and follow up data will be collected for a) functional b) neuromechanical c) cortical and d) cognitive outcomes. During walking on treadmill data will also be collected with instrumented C- MILL. C-MILL can provide gait parameters such as step length, width, frequency, speed and symmetry in addition to center of pressure for evaluation of gait and balance.

During Training Sessions: The instrumented treadmill will collect force data during training.

ELIGIBILITY:
Inclusion/exclusion criteria for TBI:

Inclusion Criteria:

Participants must:

* Be TBI survivors > 6 months post TBI
* Be able to tolerate upright standing for up to 30 minutes.
* Have joint range of motion within normal functional limits for walking as determined by study staff.
* Be between 13-35 years of age.
* Be able to follow directions and commands.
* Be able to communicate in English.
* Have stable blood pressure.
* Not been diagnosed with any cognitive (thinking) deficits.

Exclusion Criteria:

* Weight above 300lbs.
* Joint contracture or spasticity of any limb that limits normal range of motion during ambulation with assistive devices.
* Have any medical issue that prevents from supporting his/her weight (e.g. orthopedic injuries, pain, or severe spasticity).
* Have pre-existing condition that causes exercise intolerance (e.g. documented uncontrolled hypertension, coronary artery disease, irregular heart rate or rhythm, or congestive heart failure).
* Skin issues that would prevent from wearing a harness.
* Have been hospitalized for heart attack, heart surgery or acute heart failure within 3 months of enrollment in study.
* Have uncontrolled seizure disorder.
* Have uncontrolled spasticity that would interfere with walking.
* Diagnosed with cognitive (thinking) problems prior to TBI.
* Have neuromuscular or neurological issues (e.g. spinal cord injury, multiple sclerosis, or Parkinson's disease)

Inclusion/exclusion criteria for Healthy controls:

Inclusion Criteria:

Participants must:

* Be able to tolerate upright standing for up to 30 minutes.
* Have joint range of motion within normal functional limits for ambulation.
* No history of orthopedic, neuromuscular, cognitive or neurological disorders.
* Be between 13-35 years of age.
* Have stable blood pressure; no diagnosis of persistent orthostatic hypotension (blood pressure drop of more than 30 millimeters of Mercury in body weight support system).
* No diagnosed cognitive deficits.

Exclusion Criteria:

* Weight above 300lbs
* Joint contracture or spasticity of any limb that limits normal range of motion during ambulation with assistive devices.
* Any medical issue that precludes full weight bearing and ambulation (e.g. orthopedic injuries, pain, severe spasticity).
* Pressure sore that would negatively affect weight bearing, or harness fit.
* Pre-existing condition that causes exercise intolerance.(Documented uncontrolled hypertension, coronary artery disease, cardiac arrhythmia, or congestive heart failure)
* Hospitalization for heart attack, heart surgery or acute heart failure within 3 months of enrollment in study.
* Uncontrolled seizure disorder.
* Uncontrolled spasticity that would interfere with walking due to neuromuscular or neurological pathologies (e.g., Parkinson's disease, spinal cord injury, or multiple sclerosis) that will interfere with ambulation, or limit the range of motion of the lower limbs
* Diagnosed with cognitive deficits.

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2024-09-29 (Estimated); Study Completion 2024-09-29 (Estimated)

PRIMARY OUTCOMES:
Change in Dynamic Gait Index (DGI) | 5 weeks
  DGI is a measurement tool commonly used to assess dynamic balance, gait and risk for falls. It consist of a total of eight gait assessments which can be scored on a four-point ordinal scale, ranging from 0-3, where '0' indicates the lowest level of function and '3' the highest level of function, allowing for a total possible score of 24.
Change in Timed Up and Go (TUG) | 5 weeks
  TUG is a clinical test of functional gait abilities and dynamic balance. The participants will be asked to walk a distance of 3 meters from a seated position, turn around, walk back to the chair and sit back in the chair. The time taken to perform the task will be recorded using a stop watch. The TUG will be repeated multiple times. The participant may be asked to hold a plastic cup or count backwards by three from a randomly selected number while walking.
Change in Six Minute Walk | 5 weeks
  Participants walk as far as possible for 6 minutes. They walk back and forth around the cones along an unobstructed pathway of 15 meters. They will be permitted to slow down or stop as necessary. The distance covered by the participant for the 6 minutes will be recorded at an interval of every 30 seconds using a measuring wheel and stop watch.
Change in Ten Meter Walk Test | 5 weeks
  This is a walking test. I will be asked to walk as fast as I can at a safe speed for 10 meters (about 10 yards).
Change in Temporal Characteristics using pressure mat | 5 weeks
  Participants will be asked to walk about 10 meters on a pressure mat. Pressure mat (ZenoMat, Protokinetics LLC) will be used to collect gait cycle times, in order to determine inter- and intra-limb temporal characteristics.
Change in Spatial Characteristics | 5 weeks
  Participants will be asked to walk about 10 meters on a pressure mat. Pressure mat (ZenoMat, Protokinetics LLC) will be used to collect spatial parameters, in order to determine inter- and intra-limb spatial characteristics.
Change in Silver Index | 5 weeks
  Silver index using Movendo Technology platform (Movendo Technology Srl,, Italy) is an objective test that enables to predict falls by assessing static and dynamic balance. Participants will be asked to stand on the Hunova platform. Silver index includes the following tasks: stand with eyes open or eyes closed, stand when the surface is perturbed, move torso on all four sides, perform sit to stand.
Change in Cortical Activity | 5 weeks
  Cortical activity will be measured using 16 channel NIRSport 2 (NIRX Medical Technologies, LLC ), an Functional Near Infrared Spectroscopy (fNIRS) system. NIRSport 2 is a portable, non-invasive optical imaging technique to measure the cerebral hemodynamic response. fNIRS will be measure while the participants walks at a comfortable speed.
Change in Trail Making Test A and B | 5 weeks
  The task requires a subject to connect a sequence of 25 consecutive targets on a sheet of paper. Trail making Test A and B assess processing speed and executive function.
Change in Montreal Cognitive Assessment Test | 5 weeks
  30-item question to assess cognitive impairment. MoCA is used to test orientation, attention, memory, and executive function.

SECONDARY OUTCOMES:
Change in Gait Kinematics | 5 weeks
  Natural Point's optitrack camera system will be used to collect joint angles at hip, knee and ankle using reflective markers placed on the anatomical joints.
Change in Electromyography | 5 weeks
  Noraxon's surface Electromyography (EMG) wireless sensors will be used to measure the activation of tibialis anterior, soleus, vastus lateralis, rectus femoris, bicep femoris, and gastrocnemius during walking.
Change in Continuous Performance Task (CPT) | 5 weeks
  The test requires a subject to click only when presented with a target. They must refrain from clicking if they see anything other than the target. To increase the difficulty, they will be asked to click if they see another stimuli before the target. CPT assesses sustained and selective attention.
Change in C-MILL Force Data | 10 training sessions
  Force data during walking and standing will be collected during training sessions by the C-MILL

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided